CLINICAL TRIAL: NCT04962321
Title: Wellness Education Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Carrie McAdams, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-0563
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Overweight and Obesity; Eating Disorders; Depression, Anxiety
MeSH Terms: conditions — Overweight; Obesity; Feeding and Eating Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Pilot study to examine acceptability, feasibility, and explore clinical responses related to wellness behaviors and quality of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PsychoEd (Experimental): These participants are enrolled to participate in the 8-session education sessions.
  Interventions: Behavioral: Wellness Education

INTERVENTIONS:
Behavioral: Wellness Education — Psychoeducation on relationships between mood, anxiety, eating, and exercise behaviors. One one-hour session each week for 8 weeks.

SUMMARY:
Individuals suffering from depression and anxiety have an increased risk of obesity due to multiple factors such as side effects to psychotropic medications, associated appetite dysregulation, disruption of sleep, anergia leading to psychomotor retardation or inactivity, and increased stress hormones through the disruption in the hypothalamic-pituitary-adrenal (HPA) axis. Though not a causal relationship, an intimate bidirectional connection exists between the two conditions, which subsequently impacts the journey of weight loss. The impact mental health can have on weight loss is evident as concurrent depression and anxiety in individuals with obesity predicts poorer outcomes like decreased adherence and less success with weight loss interventions. Here, we will determine if delivery of psychoeducation regarding the primitive brain and model of safety in a group setting to those with obesity seeking weight loss intervention has an impact on not only psychiatric symptoms of depression and anxiety but also weight loss, eating behaviors, sleeping patterns, activity level, and health-related quality of life. This project will improve our understanding of the role of mental health and the stress response in obesity.

DETAILED DESCRIPTION:
This project will recruit subjects seeking weight loss in the Dallas Fort Worth area. A screen consisting of patient's weight and height to calculate a patient's BMI will be completed. Pre-assessment measures of anxiety, depression, eating disorder symptoms, sleep, self-efficacy, quality of life, and weight-wellness related behaviors (sleeping patterns, exercise patterns, eating patterns) will be completed before the intervention using a secure online link to RedCap. Participants will then attend eight weekly sessions of a group psychoeducational intervention. The intervention includes eight modules of various topics including the psychoeducation on the primitive brain model, motivation, goal-setting, affirmations, rewards, promoting autonomy, reducing guilt, and relapse prevention. Participants will complete homework assignments, share their work with the group to elicit feedback, and participate in guided discussions. Post-assessments will be completed 1-4 weeks and 3-5 months after the interventions is completed. These measures will determine (1) if psychological symptoms are responsive to the intervention, and (2) if clinical symptom changes related to weight and quality of life are affected.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent
* able to speak English sufficiently to understand study procedures, provide written informed consent for study participation, and complete questionnaires
* BMI > 25
* appropriate for outpatient care

Exclusion Criteria:

* medically unstable
* inpatient medical
* psychiatric inpatient
* psychiatric residential care

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Change in Physical Health Summary Scores from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For our primary measure, we will use the physical health to examine pain interference and intensity. PROMIS raw scores range from 9-50; the PROMIS T-scores have a mean of 50 with a standard deviation of 10 and where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in Mental Health Summary Scores from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For our primary measure, we will use the mental health summary score to examine anxiety, depression, and ability to participate in social roles. PROMIS raw scores range from 12-60; the PROMIS T-scores have a mean of 50 with a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in Physical Health Summary Scores from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For our primary measure, we will use the physical health to examine pain interference and intensity. PROMIS raw scores range from 9-50; the PROMIS T-scores have a mean of 50 with a standard deviation of 10 and where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in Mental Health Summary Scores from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For our primary measure, we will use the mental health summary score to examine anxiety, depression, and ability to participate in social roles. PROMIS raw scores range from 12-60; the PROMIS T-scores have a mean of 50 with a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in self-efficacy score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Generalized Self-Efficacy Scale measures how the respondent copes with daily hassles and adapts to stressful life events. Possible scores range from 10-40, with higher scores indicative of greater self-efficacy.
Change in self-efficacy score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Generalized Self-Efficacy Scale measures how the respondent copes with daily hassles and adapts to stressful life events. Possible scores range from 10-40, with higher scores indicative of greater self-efficacy.
Change in frequency of patients with eating disorders from Pre- assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Eating Disorder Screener for DSM-V (EDDS-5) screens a participant for the presence of an eating disorder. Should the screen be positive, a patient may meet criteria for an eating disorder.
Change in frequency of patients with eating disorders from Pre- assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Eating Disorder Screener for DSM-V (EDDS-5) screens a participant for the presence of an eating disorder. Should the screen be positive, a patient may meet criteria for an eating disorder.
Study components feedback score at 4 weeks after starting intervention | 4 weeks after starting intervention
  The Weight Wellness Intervention Evaluation addresses study component feedback using both a rating scales and free form written commentary. Possible scores range from 1 to 5 with higher scores indicating more positive values.
Study components feedback score at 8 weeks after starting intervention | 8 weeks after starting intervention
  The Weight Wellness Intervention Evaluation addresses study component feedback using both a rating scales and free form written commentary. Possible scores range from 1 to 5 with higher scores indicating more positive values.
Patient satisfaction score | 1-4 weeks after intervention ends
  The Weight Wellness Group Intervention Evaluation form measured patient satisfaction (the impact and value of study) with free-form verbal responses as well as a single rating scale. Possible scores range from 1 to 5 with higher scores indicating more satisfaction with the intervention.
Change in Behavioral Patterns from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Using the Wellness Pattern Questionnaire, consistency of eating, sleeping, and activity patterns are assessed. Possible scores range from 0 to 30, with higher scores reflecting more consistent scheduling for these daily behaviors.
Change in Behavioral Patterns from Pre-assessment to Post-assessment 2 | Time Frame: Baseline, 3-5 months after intervention end
  Using the Wellness Pattern Questionnaire, consistency of eating, sleeping, and activity patterns are assessed. Possible scores range from 0 to 30, with higher scores reflecting more consistent scheduling of daily behaviors.

SECONDARY OUTCOMES:
Change in weight from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Weight will be measured in pounds, percentage changed from baseline (loss or gain), and BMI.
Change in weight from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Weight will be measured in pounds, percentage changed from baseline (loss or gain), and BMI.
Change in physical function score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. T-scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in physical function score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. T-scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in depression score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in depression score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in anxiety score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in anxiety score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in fatigue score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the fatigue sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in fatigue score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the fatigue sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in sleep disturbance score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in sleep disturbance score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in ability to participate in social roles and activities score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For our secondary measure, we will examine the sleep disturbance sub-section score. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in ability to participate in social roles and activities score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For our secondary measure, we will examine the sleep disturbance sub-section score. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in pain interference score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in pain interference score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention ends
  Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 Profile, v. 2.0 Adult Profile measures the patient's perceived quality of life over the past week using various criteria. For this secondary measure, we will examine the physical function sub-section score. PROMIS raw scores for this subscale range from 4 to 20; the PROMIS T-scores have a mean 50 and a standard deviation of 10 where higher scores indicate more symptoms and less functioning. Scores up to 55 are considered to be within normal range, scores of 55-60 are indicative of mild symptoms or minor impairment, scores of 61-70 are indicative of moderate symptoms or moderate impairment, and scores greater than 71 are indicative of severe symptoms or severe impairment.
Change in ASA dietary recall data analysis of food groups from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Automated Self-administered (ASA) Dietary Recall measures the foods and beverages consumed throughout the previous day. We will compare the dietary analysis (nutrients and food groups) reported by participant on the ASA Dietary Recall.
Change in ASA dietary recall data analysis of food groups from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention end
  Automated Self-administered (ASA) Dietary Recall measures the foods and beverages consumed throughout the previous day. We will compare the dietary analysis (nutrients and food groups) reported by participant on the ASA Dietary Recall.
Change in sleep pattern score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Using the Wellness Patterns Questionnaire, effort and ability to keep a regular sleep schedule are assessed. Possible scores range from 0 to 7, with higher scores indicating a more regular sleep pattern.
Change in sleep pattern score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention end
  Using the Wellness Patterns Questionnaire, effort and ability to keep a regular sleep schedule are assessed. Possible scores range from 0 to 7, with higher scores indicating a more regular sleep pattern.
Change in eating pattern score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Using the Wellness Patterns Questionnaire, eating effort and ability to keep a regular eating pattern are assessed. Possible scores range from 0 to 16, with higher scores suggesting more consistent eating patterns.
Change in eating pattern score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention end
  Using the Wellness Patterns Questionnaire, effort and ability to keep a regular eating pattern are assessed. Possible scores range from 0 to 16, with higher scores suggesting more consistent eating patterns.
Change in activity score from Pre-assessment to Post-assessment 1 | Baseline, 1-4 weeks after intervention ends
  Using the Wellness Patterns Questionnaire, consistency of exercise and activity patterns is assessed. Possible scores range from 0 to 7, with higher scores reflecting more consistent engagement in exercise.
Change in activity score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention end
  Using the Wellness Patterns Questionnaire, consistency of exercise and activity patterns is assessed. Possible scores range from 0 to 7, with higher scores reflecting more consistent engagement in exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie J McAdams, MD PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No